CLINICAL TRIAL: NCT05249842
Title: Respiratory Function 3 Months After Hospital Discharge in Critically Ill COVID-19 Patients
Status: Completed | Type: Observational
Sponsor: Hospital Sao Domingos (Other)
Responsible Party: Principal Investigator, José Raimundo Araujo de Azevedo, ICU Coordinator, Hospital Sao Domingos
Other Study IDs: 53
Record Dates: First submitted 2022-02-19; First posted 2022-02-22 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: COVID-19
Keywords: COVID-19; Critical Care; Survivors; Pulmonary function test; Physical component summary
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Respiratory function 3 months after hospital discharge in critically ill COVID-19 patients: All critically ill adult patients admitted to the ICU with confirmed diagnosis of COVID-19 were submitted at least 3 months after hospital discharge to spirometry (FVC, FEV1, FEV1 /;FVC and FEF 25-75%), the 6-minute walk test (6MWT) and evaluation of the physical component summary (PCS) of the SF-36 quality of life instrument.
  Interventions: Diagnostic Test: Spirometric evaluation; Diagnostic Test: Physical component summary; Diagnostic Test: 6MWT

INTERVENTIONS:
Diagnostic Test: Spirometric evaluation — Evaluation of: forced vital capacity (FVC),, FEV1', FEV 1/FVC, FEF 25-75
Diagnostic Test: Physical component summary — Evaluation of the physical component summary of SF-36 quality of life
Diagnostic Test: 6MWT — 6 minute walk test

SUMMARY:
The objective of this single-center retrospective observational study is to describe spirometric abnormalities and their impact on 6-minute walk test (6MWT) and the physical component summary (PCS) of the SF-36 quality of life instrument.at least 3 months later discharge hospital.

DETAILED DESCRIPTION:
Background: The COVID-19 pandemic has already affected more than 400 million people worldwide and resulted in at least 6 million deaths. The disease has also resulted in a growing population of individuals, with both physical and mental sequelae. Pulmonary sequelae have been the subject of several studies because the lung is the main target organ of the disease. However, there is still unknown data about the pulmonary manifestations and their spirometric patterns after a critical illness and also its consequences in quality of life.

Purpose: Up to 20% of COVID-19 patients develop severe forms of the disease and require ICU admission. Most of these patients at hospital discharge still have several limitations that impact on quality of life. Some studies have analyzed pulmonary functional alterations after a variable period of time and have found results that vary from the absence of functional alterations to restrictive and diffusion impairment. Few studies have analyzed changes in small airways, and those that have evaluated have found no changes. The objective of this single-center retrospective observational study is to describe spirometric abnormalities and their impact on 6-minute walk test (6MWT) and the physical component summary (PCS) of the SF-36 quality of life instrument.at least 3 months later discharge hospital.

Primary outcome: To describe spirometric patterns associated to severe COVID-19 survivors at least 3 months after hospital discharge.

Secondary outcomes: Correlate the results of the spirometric evaluation with the 6-minute walk test (6MWT) and the physical component summary (PCS) of the SF-36 quality of life instrument.

Methods: An observational retrospective study will be conducted, including all 18 years and older patients with severe COVID-19, confirmed by real-time reverse transcriptase-polymerase chain reaction., admitted to a 35- bed intensive care unit of a tertiary hospital from April 2020 to October 2021. Pediatric, pregnant or breastfeeding women and palliative care patients as well as chronic obstructive pulmonary disease and symptomatic asthmatic patients will be excluded. Population is estimated at 60 patients. Data collecting will be finished in February 2022. Patients routinely are assessed after at least 3 months after hospital discharge in our multidisciplinary follow-up clinic. A trained research team will routinely apply the 6 minute walk test (6MWT), a Pulmonary Function Test (PFT) and Short Form Health Survey 36 (SF-36) physical component summary (PCS) of SF-36

ELIGIBILITY:
Inclusion Criteria

* All 18 years and older patients with severe COVID-19, confirmed by real-time reverse transcriptase-polymerase chain reaction., admitted to a 15- bed intensive care unit of a tertiary hospital from April 2020 to October 2021.

Exclusion criteria

* < 18 years old
* Pregnant
* Breastfeeding
* Chronic pulmonary obstructive disease
* Symptomatic asthma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with confirmed COVID-19 admitted to the ICU requiring non-invasive or invasive respiratory support
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Forced vital capacity (FVC) | 3 months after hospital discharge
  Forced vital capacity (FVC) is the volume of air that can forcibly be blown out after full inspiration, Measured in liters. Normal value > 80% of predicted for age, sex, heigth and ethnicity
Forced expiratory volume in 1 second (FEV1) | 3 months after hospital discharge
  FEV1 is the volume of air that can forcibly be blown out in first 1 second, after full inspiration. Measured in liters. Normal value > 80%. of predicted for age, heigth and ethnicity.
FEV1 / FVC Ratio | 3 months after hospital discharge
  Represents the proportion of vital capacity that the patients are able to expire in the first second of forced expiration (FEV1) to the full, forced vital capacity (FVC). The result of this ratio is expressed as FEV1%. Normal values are > 75%.of predicted that depend on age, sex, height, and ethnicity
Forced mid-expiratory flow (FEF25-75%) | 3 months after hospital discharge
  Defined as the mean forced expiratory flow during the middle half of the FVC . Normal value > 65% of predictedf for age, sex, heigth and ethnicity

SECONDARY OUTCOMES:
Physical Component Summary (PCS) of Short Form- 36 (SF-36) Instrument | 3 months after hospital discharge
  PCS is composed of four scales assessing physical function, role limitations caused by physical problems, bodly pain and general health. The result scale ranges from 0 to 100, with 0 being the worst result and 100 the best.
6 Minute Walk Test | 3 months after hospital discharge
  The patient is placed on a flat, rigid area 30 meters long and instructed to walk the longest tolerable distance for 6 minutes. Measured in meters. The result is given as a percentage of the normal predicted value for age, sex, height and weight calculated by the Enright and Sherril equation.

CONTACTS AND LOCATIONS:
Overall Officials: JOAQUIM LOBATO, MD, Principal Investigator — Hospital Sao Domingos
Locations (1):
- Hospital Sao Domingos, São Luís, Maranhão, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang Y, Tan C, Wu J, Chen M, Wang Z, Luo L, Zhou X, Liu X, Huang X, Yuan S, Chen C, Gao F, Huang J, Shan H, Liu J. Impact of coronavirus disease 2019 on pulmonary function in early convalescence phase. Respir Res. 2020 Jun 29;21(1):163. doi: 10.1186/s12931-020-01429-6. PMID 32600344
- [Background] Graham BL, Steenbruggen I, Miller MR, Barjaktarevic IZ, Cooper BG, Hall GL, Hallstrand TS, Kaminsky DA, McCarthy K, McCormack MC, Oropez CE, Rosenfeld M, Stanojevic S, Swanney MP, Thompson BR. Standardization of Spirometry 2019 Update. An Official American Thoracic Society and European Respiratory Society Technical Statement. Am J Respir Crit Care Med. 2019 Oct 15;200(8):e70-e88. doi: 10.1164/rccm.201908-1590ST. PMID 31613151
- [Result] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Result] Hui DS, Joynt GM, Wong KT, Gomersall CD, Li TS, Antonio G, Ko FW, Chan MC, Chan DP, Tong MW, Rainer TH, Ahuja AT, Cockram CS, Sung JJ. Impact of severe acute respiratory syndrome (SARS) on pulmonary function, functional capacity and quality of life in a cohort of survivors. Thorax. 2005 May;60(5):401-9. doi: 10.1136/thx.2004.030205. PMID 15860716
- [Result] Frija-Masson J, Debray MP, Gilbert M, Lescure FX, Travert F, Borie R, Khalil A, Crestani B, d'Ortho MP, Bancal C. Functional characteristics of patients with SARS-CoV-2 pneumonia at 30 days post-infection. Eur Respir J. 2020 Aug 6;56(2):2001754. doi: 10.1183/13993003.01754-2020. Print 2020 Aug. PMID 32554533
- [Result] Li X, Wang C, Kou S, Luo P, Zhao M, Yu K. Lung ventilation function characteristics of survivors from severe COVID-19: a prospective study. Crit Care. 2020 Jun 6;24(1):300. doi: 10.1186/s13054-020-02992-6. No abstract available. PMID 32505211
- [Result] Mo X, Jian W, Su Z, Chen M, Peng H, Peng P, Lei C, Chen R, Zhong N, Li S. Abnormal pulmonary function in COVID-19 patients at time of hospital discharge. Eur Respir J. 2020 Jun 18;55(6):2001217. doi: 10.1183/13993003.01217-2020. Print 2020 Jun. PMID 32381497
- [Result] You J, Zhang L, Ni-Jia-Ti MY, Zhang J, Hu F, Chen L, Dong Y, Yang K, Zhang B, Zhang S. Anormal pulmonary function and residual CT abnormalities in rehabilitating COVID-19 patients after discharge. J Infect. 2020 Aug;81(2):e150-e152. doi: 10.1016/j.jinf.2020.06.003. Epub 2020 Jun 5. No abstract available. PMID 32512021
- [Result] Zhao YM, Shang YM, Song WB, Li QQ, Xie H, Xu QF, Jia JL, Li LM, Mao HL, Zhou XM, Luo H, Gao YF, Xu AG. Follow-up study of the pulmonary function and related physiological characteristics of COVID-19 survivors three months after recovery. EClinicalMedicine. 2020 Aug;25:100463. doi: 10.1016/j.eclinm.2020.100463. Epub 2020 Jul 15. PMID 32838236
- [Result] Ngai JC, Ko FW, Ng SS, To KW, Tong M, Hui DS. The long-term impact of severe acute respiratory syndrome on pulmonary function, exercise capacity and health status. Respirology. 2010 Apr;15(3):543-50. doi: 10.1111/j.1440-1843.2010.01720.x. Epub 2010 Mar 19. PMID 20337995
- [Result] Lindahl A, Reijula J, Malmberg LP, Aro M, Vasankari T, Makela MJ. Small airway function in Finnish COVID-19 survivors. Respir Res. 2021 Aug 26;22(1):237. doi: 10.1186/s12931-021-01830-9. PMID 34446020
- [Result] Polese J, Sant'Ana L, Moulaz IR, Lara IC, Bernardi JM, Lima MD, Turini EAS, Silveira GC, Duarte S, Mill JG. Pulmonary function evaluation after hospital discharge of patients with severe COVID-19. Clinics (Sao Paulo). 2021 Jun 28;76:e2848. doi: 10.6061/clinics/2021/e2848. eCollection 2021. PMID 34190851
- [Result] Torres-Castro R, Vasconcello-Castillo L, Alsina-Restoy X, Solis-Navarro L, Burgos F, Puppo H, Vilaro J. Respiratory function in patients post-infection by COVID-19: a systematic review and meta-analysis. Pulmonology. 2021 Jul-Aug;27(4):328-337. doi: 10.1016/j.pulmoe.2020.10.013. Epub 2020 Nov 25. PMID 33262076